CLINICAL TRIAL: NCT01834651
Title: A Phase II Study of Cabozantinib (XL184) Therapy in Castrate Resistant Prostate Cancer (CRPC) With Visceral Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Edwin Posadas, MD (Other)
Responsible Party: Sponsor-Investigator, Edwin Posadas, MD, Medical Director, Urologic Oncology Program, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL184-IST20
Record Dates: First submitted 2013-04-01; First posted 2013-04-18 (Estimated); Results first posted 2017-09-27 (Actual); Last update posted 2017-09-27 (Actual); Status verified 2017-08

CONDITIONS: Prostate Cancer
Keywords: liver metastasis; lung metastasis; metastatic castrate-resistant; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cabozantinib) (Experimental): Cabozantinib 60mg orally daily until disease progression
  Interventions: Drug: Cabozantinib

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib 60 mg daily (oral). Subjects may continue to receive study treatment until they experience unacceptable drug-related toxicity or disease progression.
  Other Names: XL184

SUMMARY:
This research study is being done to measure the clinical benefit associated with cabozantinib (XL184) in men who have prostate cancer that has spread to visceral organs (organs other than bone or lymph nodes) and no longer responds to initial hormonal (castration) therapy. This type of prostate cancer is called metastatic, castrate-resistant prostate cancer.

DETAILED DESCRIPTION:
Cabozantinib (XL184), a multi-targeted tyrosine kinase inhibitor, has demonstrated a powerful clinical phenotype in men with metastatic castrate resistant prostate cancer (mCRPC) both before and after chemotherapy. This phenotype consists of rapid reduction in pain (when present) and improvement in bone scans that may or may not be accompanied by decrease in serum prostate specific antigen (PSA) concentrations. In previous studies of cabozantinib in advanced prostate cancer, patients with visceral disease have been excluded. Hence, this protocol creates a unique opportunity to define the activity of this disease in the population of men with visceral disease - a marker for poorer prognosis in mCRPC.

Primary Objectives:

- To assess the clinical benefit (complete response + partial response + stable disease) of cabozantinib in patients with mCRPC with visceral metastases.

Secondary Objectives:

* To assess the impact of cabozantinib on numbers live circulating tumor cells (CTCs) using NanoVelcro Chips
* To test the feasibility of measuring variation in gene expression in circulating tumor cells (CTCs) in response to therapy.
* To determine if there is an impact of cabozantinib on live circulating tumor cell (CTC) number and patterns of gene expression.
* To measure the impact of cabozantinib on serum HGF (hepatocyte growth factor) and VEGF (vascular endothelial growth factor) levels in men with metastatic, castration-resistant prostate cancer (mCRPC).
* To assess the safety and tolerability of lower doses (i.e. doses below 100 mg daily) of cabozantinib in mCRPC with visceral involvement.
* To collect blood, urine, tissue, and plasma which may be used determine if there are germline genetic variations that correlate with toxicity.
* To pilot correlations between molecular content between circulating tumor cells (CTCs), large oncosomes, and tumor tissue.

ELIGIBILITY:
KEY INCLUSION CRITERIA

- mCRPC that includes visceral disease. Visceral metastatic disease is defined as solid organ infiltration that is not bone or lymph node metastases.

KEY EXCLUSION CRITERIA

* Recent history (<6 months) of gastrointestinal hemorrhage requiring blood transfusion.
* Tumor involvement in the intestinal lining which the treating physician deems at risk for perforation with rapid tumor response.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-04-30 (Actual); Primary Completion 2016-07-18 (Actual); Study Completion 2016-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Posadas, MD FACP, Principal Investigator — Cedars-Sinai Medical Center Samuel Oschin Comprehensive Cancer Institute
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Cabozantinib)
Started | 17
Completed | 16 (Evaluable for primary outcome assessment at 12 weeks)
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Cabozantinib)
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 65 [50 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate From Cabozantinib (XL184)
Description: Clinical benefit rate is defined as the combination of complete response, partial response, and stable disease as defined by modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as assessed by CT imaging and Prostate Cancer Working Group 2 (PCWG2) criteria.
  Complete response (CR) defined as disappearance of all target lesions; Partial response (PR) >=30% decrease in som of diameters of target lesions (taking as reference the baseline), and stable disease, neither sufficient shrinkage to qualify for PR nor increase to qualify for progressive disease.
Time Frame: Baseline to 12 weeks after starting therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cabozantinib)
Number analyzed (Participants) | 16
Participants | 10

2. Secondary Outcome: Change in Number of Circulating Tumor Cells (CTC) in Response to Cabozantinib
Description: Change in number of CTC from baseline at 12 weeks
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: CTCs/7.5 ml
Arm/Group | Treatment (Cabozantinib)
Number analyzed (Participants) | 14
CTCs/7.5 ml | 53.2 (217.8)

3. Secondary Outcome: Number of Patients With NanoVelcro Appropriate for RNA in Circulating Tumor Cells
Description: This is to provide a measure of feasibility using NanoVelcro to measure RNA in circulating tumor cells (CTC)
Time Frame: 12 weeks
Population: There were 16 patients evaluable for this outcome (1 patient did not have RECIST measurable disease)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cabozantinib)
Number analyzed (Participants) | 16
Participants | 16

4. Secondary Outcome: Change in Levels of Serum Hepatocyte Growth Factor (HGF) and Vascular Endothelial Growth Factor (VEGF) Concentration
Description: Mean change from baseline in levels of HGF and VEGF
Time Frame: 12 weeks
Population: HGF was evaluable in 16 patients who had viable research samples. VEGF was evaluable in 15 patients who had viable research samples.
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Treatment (Cabozantinib) HGF Levels: Cabozantinib 60mg orally daily until disease progression
  Cabozantinib: Cabozantinib 60 mg daily (oral). Subjects may continue to receive study treatment until they experience unacceptable drug-related toxicity or disease progression.
- Treatment (Cabozantinib) VEGF Levels: Carbozantinib 60mg
Arm/Group | Treatment (Cabozantinib) HGF Levels | Treatment (Cabozantinib) VEGF Levels
Number analyzed (Participants) | 16 | 15
pg/ml | -322.96 (1981.19) | 191.1 (302.1)

5. Secondary Outcome: Number of Participants With Grade 3/4 Adverse Events Related to Cabozantinib as Assessed Using CTCAE (v.4)
Description: Each cycle is 28 days. Safety and tolerability was defined as related grade 3-4 AEs of doses of cabozantinib below 100 mg daily using common terminology criteria for adverse events (CTCAE)
Time Frame: Every 2 weeks for first 3 Cycles and every 4 weeks thereafter for an expected average of 28 weeks.
Population: All patients
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cabozantinib)
Number analyzed (Participants) | 17
Participants
  AST increased | 4
  Alkaline phosphatase increased | 2
  Anemia | 1
  Corneal Epithelial Defect | 1
  Dehydration | 1
  Diarrhea | 1
  GGT increased | 1
  Hematuria | 1
  Hypertension | 1
  Hyponatremia | 2
  Lipase increased | 2
  Lymphocyte count decreased | 3
  Palmar-Plantar Erythrodysesthesia | 1
  Rectal Fistula | 1

6. Secondary Outcome: Number of Patients With Evaluable Protein Content of Large Oncosomes From Baseline to First Documented Progression or Date of Death
Description: This is a feasibility outcome to assess ability to measure protein content in large oncosomes in this population.
Time Frame: From baseline until the date of first documented progression or date of death from any cause, whichever comes first, assessed for an expected average of 28 weeks.
Population: Only 12 samples were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cabozantinib)
Number analyzed (Participants) | 12
Participants | 12

ADVERSE EVENTS:
Time Frame: From signed consent up to 30 days after last treatment
Description: Attributions and ratings completed by Investigators as per CTCAE
Arm/Group | Treatment (Cabozantinib)
Serious Adverse Events (participants affected / at risk) | 14/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Cabozantinib) (N=17)
Anemia (Blood and lymphatic system disorders) | 3
Chest Pain- Cardiac (Cardiac disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Confusion (Psychiatric disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fever (General disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Keratitis (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Rectal fistula (Gastrointestinal disorders) | 1
Retinal detachment (Eye disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Cabozantinib) (N=17)
ALT increased (Investigations) | 17
AST increased (Investigations) | 15
Abdominal pain (Gastrointestinal disorders) | 4
Activated PTT prolonged (Investigations) | 2
Alkaline Phosphatase increased (Investigations) | 11
Allergic Reaction (Immune system disorders) | 1
Allergic Rhinitis (Immune system disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anasarca (Skin and subcutaneous tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 8
Anorexia (Metabolism and nutrition disorders) | 9
Anxiety (Psychiatric disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bacterial Overgrowth (Reproductive system and breast disorders) | 1
Blepharitis (Eye disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Blood Bilirubin Increased (Investigations) | 4
Blurred Vision (Eye disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 2
Cataract (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Corneal Epithelial Defect (Eye disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine Increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 10
Diplopia (Eye disorders) | 1
Dizziness (Nervous system disorders) | 2
Dry eye (Eye disorders) | 3
Dry mouth (Gastrointestinal disorders) | 4
Dry nose (Skin and subcutaneous tissue disorders) | 1
Dysguesia (Nervous system disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Edema limbs (General disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Inflamed eyelids (Eye disorders) | 1
Eye Pain (Eye disorders) | 1
Facial Rash (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 9
Fecal Incontinence (Gastrointestinal disorders) | 1
Fever (General disorders) | 4
Flatulence (Gastrointestinal disorders) | 2
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 4
GGT Increased (Investigations) | 10
Genital Edema (Reproductive system and breast disorders) | 1
Gynecomastia (Reproductive system and breast disorders) | 2
Hair Color Change (Skin and subcutaneous tissue disorders) | 3
Hematuria (Renal and urinary disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 10
Hot Cold (General disorders) | 1
Hot Flashes (General disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 10
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 10
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hypotension (Vascular disorders) | 2
Hypothyroidism (Metabolism and nutrition disorders) | 3
Insomnia (Psychiatric disorders) | 1
Keratitis (Eye disorders) | 1
Lipase Increased (Investigations) | 3
Localized edema - bilateral leg (General disorders) | 1
Lymphocyte Count Decreased (Blood and lymphatic system disorders) | 11
Mucositis Oral (Gastrointestinal disorders) | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Nail Changes (Skin and subcutaneous tissue disorders) | 1
Nasal Discharge (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Nervous system disorders other, T5 - T9 co (Nervous system disorders) | 1
Neutrophil Count Decreased (Investigations) | 3
Oculomotor Nerve Disorder (3rd Nervepalsy) (Nervous system disorders) | 1
Osteonecrosis of Jaw (Musculoskeletal and connective tissue disorders) | 1
Pain (General disorders) | 1
Pain (Pain in Jaw) (General disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 13
Paresthesia (Nervous system disorders) | 1
Paronychia (Infections and infestations) | 1
Platelet Count Decreased (Investigations) | 8
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Presyncope (Nervous system disorders) | 1
Psychiatric disorders - Other, Nightmares (Psychiatric disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rectal Fistula (Gastrointestinal disorders) | 2
Right Foot Drop (Musculoskeletal and connective tissue disorders) | 1
Scalp Follicullitos (Skin and subcutaneous tissue disorders) | 1
Serum Amylase Increased (Investigations) | 3
Sinus Tachycardia (Cardiac disorders) | 2
Skin Friable (Skin and subcutaneous tissue disorders) | 1
Skin Induration (Skin and subcutaneous tissue disorders) | 1
Skin discoloration (Skin and subcutaneous tissue disorders) | 1
Somnolence (Psychiatric disorders) | 1
Stool Color Change (Gastrointestinal disorders) | 1
Surgical and medical procedures- Herniorrhaphy (Gastrointestinal disorders) | 1
TMJ (Nervous system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Urinary Tract Infection (Infections and infestations) | 1
Urinary Tract Obstruction (Renal and urinary disorders) | 2
Vision Change (Eye disorders) | 1
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Intermittent) (Gastrointestinal disorders) | 3
Watering Eyes (Eye disorders) | 1
Weakness (General disorders) | 1
Weight Loss (Investigations) | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
White Blood Cell Decreased (Investigations) | 11
hyperglycemia (Metabolism and nutrition disorders) | 1
proteinuria (Metabolism and nutrition disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No